CLINICAL TRIAL: NCT04773951
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Recombinant Humanized Monoclonal Antibody Specific to B- and T- Lymphocyte Attenuator, BTLA (JS004) Injection in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of JS004 in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMO-JS004-I-CT01
Record Dates: First submitted 2021-01-17; First posted 2021-02-26 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-01

CONDITIONS: Melanoma; Renal Carcinoma; Urothelial Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Carcinoma, Transitional Cell | interventions — BTLA protein, human; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation and extension group (Experimental): 1. JS004 dose escalation: 1mg/kg, IV Q3W; 3mg/kg, IV Q3W; 10mg/kg, IV Q3W;
  2. JS004 dose extension: 3mg/kg, IV Q3W; 200mg, IV Q3W;
  3. JS004+Toripalimab Injection dose escalation: JS004 100mg+Toripalimab Injection 240mg, IV Q3W; JS004 200mg+Toripalimab Injection 240mg, IV Q3W;
  4. JS004+Toripalimab Injection dose extension: JS004 100mg+Toripalimab Injection 240mg, IV Q3W or JS004 200mg+Toripalimab Injection 240mg, IV Q3W，to be determined.
  Interventions: Biological: JS004, a recombinant humanized, IgG4κ monoclonal antibody (mAb) specific to B- and T-lymphocyte attenuator (BTLA); Toripalimab Injection

INTERVENTIONS:
Biological: JS004, a recombinant humanized, IgG4κ monoclonal antibody (mAb) specific to B- and T-lymphocyte attenuator (BTLA); Toripalimab Injection — Biological: JS004, Intravenous infusion; Toripalimab Injection, Intravenous infusion

SUMMARY:
An open-label, dose-escalation, phase I clinical study to evaluate the safety and tolerability of JS004 injection in the patients with advanced solid tumors who have failure in standard of care and are unable to tolerate standard of care and/or have no available standard of care. The study is divided into screening period, treatment period, and follow-up period.

1. Screening period: Subjects will be included in the screening period after signing the informed consent form (ICF). The screening period is up to 28 days, subjects will enter the study treatment period if they meet all the inclusion criteria and none of exclusion criterion.
2. Treatment period: Subjects will be allocated to the designated dose group to receive corresponding treatment in accordance with the progress of study. Subjects in dose escalation phase will receive DLT observation at first, and upon completion of DLT observation, the subjects will continue their administration at the original dose if they are tolerated as judged by investigator, until progression of disease, intolerable toxicity or other reasons specified in the protocol. Subjects in the dose extension phase receive appropriate study treatment until disease progression, intolerance of toxicity, or other causes specified in the protocol occur. Response evaluation criteria in solid tumors (RECIST v1.1) will be used for efficacy evaluation every 9 weeks (±7 days) in the first year and every 12 weeks (±7 days) in the 2nd year and thereafter.
3. Follow-up period: A safety follow-up visit is required 30 days (±7 days) after the last dose of study drug or before the initiation of new antitumor therapy. If the new antitumor therapy has not been initiated, additional safety follow-up should be completed 90 days (±7 days) after the last dose as far as possible.

ELIGIBILITY:
Inclusion Criteria:

Only the patients meeting the following criteria are eligible to participate in the study:

1. Voluntarily signed written informed consent form;
2. Age ≥18 and ≤70 years at the time of signing informed consent form, male or female;
3. Life expectancy ≥ 3 months;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1;
5. Patients with histologically or cytologically confirmed advanced solid tumors: patients with advanced solid tumors who have failure in standard of care, cannot tolerate standard of care, refuse and/or have no standard of care (melanoma, renal carcinoma and urothelial carcinoma);
6. At least one measurable lesion as target lesion (RECIST v1.1);
7. Agree to provide tumor tissue specimen ( fresh biopsied sample before treatment should be provided as far as possible, the archived sample within two years is acceptable for the patients who cannot provide fresh biopsied sample before treatment);
8. Adequate organ function as indicated by the laboratory results during the screening period;
9. Use of effective contraceptive methods during the study for male subjects of reproduction ability or female subjects of childbearing potential, and continuation of contraception for 6 months after the end of treatment;
10. Good compliance, cooperation with follow-up.

Exclusion Criteria

Patients will be excluded from the study when they have any of the following conditions:

1. History of malignant tumors other than the disease investigated in the past 5 years, however, except for the malignant tumors that can be expected to be cured after treatment;
2. Having received systematic antitumor therapy, or local antitumor therapy, or treatment with clinically investigational medication or device within 4 weeks prior to the first dose of study drug;
3. Having received immunotherapy within 4 weeks prior to first dose of study drug;
4. Previously treated with anti-BTLA or anti-HVEM antibody;
5. Adverse reaction induced by previous therapy having not recovered to CTCAE (version 5.0) grade 1 or better;
6. Having previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
7. Having central nervous system metastases and/or cancerous meningitis;
8. Having or suspected to have active autoimmune disease;
9. Having hepatitis and liver cirrhosis;
10. Massive hydrothorax or ascites with clinical symptoms or requiring symptomatic treatment;
11. Having severe cerebro- and cardiovascular diseases;
12. Having pulmonary disease;
13. Having active infection requiring systemic treatment;
14. Positive result for human immunodeficiency virus (HIV) antibody;
15. Active hepatitis B or C;
16. Known active tuberculosis (TB);
17. Use of systemic corticosteroids 14 days prior to the first dose of study drug;
18. Use of broad-spectrum antibiotics that may affect the change of intestinal flora within 14 days prior to the first dose of study drug;
19. Vaccination of live vaccine within 4 weeks prior to the first dose of study drug;
20. Having received major surgery within 4 weeks prior to the first dose of study drug;
21. History of anti-psychotics abuse and unable to abstain, or with a history of mental disorder;
22. Pregnant or breast-feeding women;
23. Known allergy to JS004 and its components;
24. Other severe, acute or chronic medical conditions or mental diseases or laboratory abnormalities possibly increasing relevant risks in participation in the study or possibly interfering with the interpretation of study results as judged by investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of JS004 injection alone and in combination with Toripalimab in patients with advanced solid tumors. | 2 years
  Including incidence of dose limiting toxicity (DLT); incidence and severity of adverse event (AE), serious adverse event (SAE) and immune related adverse event (irAE); laboratory results with clinical significance and other tests with abnormal results.
Determine the maximum tolerated dose (MTD)/recommended extended dose (RDE) of JS004 injection monotherapy and combination with Toripalimab in patients with advanced solid tumors. | 2 years
  The maximum tolerated dose (MTD) is defined as the maximum dose at which <1/3 subjects experience any DLTs and at least 6 evaluable subjects are required at each dose level.

SECONDARY OUTCOMES:
To preliminarily evaluate the efficacy of JS004 injection as a single drug and combined with Toripalimab. | 2 years
  Objective response rate (ORR), duration of response (DOR), disease control rate (DCR), time to response (TTR), progression-free survival (PFS) in accordance with RECIST 1.1 and overall survival (OS).
To evaluate the pharmacokinetic profile of JS004 Injection as a single drug and combined with Toripalimab. | 2 years
  Drug concentration in individual subject at different time points after administration.
To evaluate the pharmacokinetic profile of JS004 Injection as a single drug and combined with Toripalimab. | 2 years
  Peak concentration (Cmax)
To evaluate the pharmacokinetic profile of JS004 Injection as a single drug and combined with Toripalimab. | 2 years
  Time to peak (Tmax)
To evaluate the pharmacokinetic profile of JS004 Injection as a single drug and combined with Toripalimab. | 2 years
  Area under the serum concentration-time curve (AUC0-t and AUC0-∞)
To evaluate the pharmacokinetic profile of JS004 Injection as a single drug and combined with Toripalimab. | 2 years
  Clearance (CL)
To evaluate the pharmacokinetic profile of JS004 Injection as a single drug and combined with Toripalimab. | 2 years
  Volume of distribution under steady state (Vss)
To evaluate the pharmacokinetic profile of JS004 Injection as a single drug and combined with Toripalimab. | 2 years
  Mean retention time (MRT)
To evaluate the pharmacokinetic profile of JS004 Injection as a single drug and combined with Toripalimab. | 2 years
  Elimination half-life (t1/2)

OTHER OUTCOMES:
To exploratively evaluate the antitumor activity of JS004 injection as a single drug and combined with Toripalimab using iRECIST (2017). | 2 years
  Objective response rate (ORR), duration of response (DOR), disease control rate (DCR) and progression-free survival (PFS) evaluated in accordance with iRECIST(2017).
To explore the pharmacodynamic profile of JS004 injection. | 2 years
  Pharmacodynamic variables related with targets: lymphocyte subpopulation, receptor occupancy.
To explore the correlation of relevant biomarkers with clinical efficacy. | 2 years
  Tumor tissue related biomarker: including but not limited to HVEM and PD-L1; density of CD8 positive tumor infiltrating immune cells; tumor tissue whole exon sequencing (WES); Peripheral blood related biomarker: cytokine; surface receptor on immune cell (including PD-1，HVEM, CTLA-4, CD112R, TIM-3, ICOS, CX3CR1, CD183, CD103).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (11):
- China (11):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Tumor Hospital affiliated to Harbin Medical University, Harbin, Heilongjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Run Run Shaw Hospital affiliated to Zhejiang University Medical College, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan